CLINICAL TRIAL: NCT06541899
Title: Safety and Efficacy of Cryolipolysis Clinical Protocols
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indústria Brasileira Equipamentos Médicos - IBRAMED (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ibramed_01_2024_V1
Record Dates: First submitted 2024-07-31; First posted 2024-08-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Fat Loss
Keywords: Fat Loss; Weight Loss; Cryolipolysis
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group 1 - 360° M applicator, abdominal (Experimental): Group 1: 360° M applicator - Abdominal region
  Interventions: Device: Polarys Cryolipolysis
- Group 2 - 360° G applicator, abdominal (Experimental): Group 2: 360° G applicator - Abdominal region
  Interventions: Device: Polarys Cryolipolysis
- Group 3 - flanks (Experimental): Group 3: Plate applicator - Flank region
  Interventions: Device: Polarys Cryolipolysis

INTERVENTIONS:
Device: Polarys Cryolipolysis — The procedure will take place in a session lasting a maximum of 60 minutes, which may vary depending on the amount of fat in the area and the type of applicator chosen (with or without vacuum). The patient will be comfortably positioned, in a position that facilitates suction/fixation of the applicator. An antifreeze membrane will be applied correctly to the skin, avoiding wrinkles. The marked skin area will be positioned in the center of the membrane. The applicator will be positioned in the treatment area at 90° to the skin and will activate the START.
  Other Names: Cryolipolysis

SUMMARY:
A single-arm, multicenter interventional clinical study will be conducted. The objective is to evaluate the safety and efficacy of the cryolipolysis technique. Approximately 372 participants will be included. After analyzing the items listed above, the participants in each study will be divided into 3 distinct intervention groups. The individuals included in the study will undergo anamnesis and data collection.

DETAILED DESCRIPTION:
The participants in each study will be divided into 3 distinct intervention groups (Grupo 1: aplicador 360° M - Região abdominal; Grupo 2: aplicador 360° G - Região abdominal; Grupo 3: aplicador de placas - Região dos flancos). After analyzing the inclusion and exclusion criteria of this study, the individuals included in the study will undergo anamnesis and data collection after the procedure and 6 weeks and 20 weeks after: photographic capture, bioimpedance, perimetry, adipometry and ultrasound imaging of the treated area, in addition to a pain and patient satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* The participant (healthy volunteer) who has read and signed the informed consent form for the study.
* Male or female ≥ 22 years and ≤ 65 years of age.
* Subjects with a body mass index (BMI) of 30 or less and who have a greater volume of adipose tissue in the abdomen (except precordial region) and flanks.
* Subject has not changed in weight more than 5% of body weight in the previous month.
* Subject agrees to maintain his/her weight (i.e., within 5%) by not making major changes in his/her diet or exercise routine during the study.
* Subject agrees to have photographs taken of the treatment area(s) during the scheduled periods.

Exclusion Criteria:

* Diabetes mellitus or need to administer or known history of subcutaneous injections in the area of intended treatment (e.g. heparin, insulin) in the last month;
* Metabolic and/or liver diseases that compromise vitamin metabolism;
* Being pregnant or planning to become pregnant during the study period (within the next 8 months);
* Being breast-feeding or having breast-fed in the last 6 months;
* Having a known sensitivity to cold, such as cold urticaria, Raynaud's disease, chilblains (pernio) or any known condition with a response to cold exposure that limits blood flow to the skin;
* Irritated skin or presence of dermatitis;
* Keloids or propensity for keloids in the area to be treated;
* Having a history of hernia in the area(s) to be treated.
* Any dermatological conditions, such as moderate to excessive skin laxity, or scarring at the location of the treatment sites that may interfere with treatment or evaluation (stretch marks are not an exclusion);
* Have a history of a bleeding disorder or are taking any medications that, in the opinion of the investigator, may increase the risk of bruising;
* Recent surgery at the treatment site;
* Regular use of anti-inflammatory medications;
* Are taking or have taken any pills or dietary supplements within the past month.
* Invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the intended treatment area;
* Implanted electronic devices (e.g., pacemaker);
* Are currently enrolled in a clinical trial of any unapproved investigational drug or device.
* Any other condition or laboratory value that could, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Ocurrence of adverse events after de procedure assessed by clinical evaluation | After de procedure and 6 and 20 weeks after
  Adverse events such as erythema, pain, edema or any other event that occurs in correlation with the treatment, through monitoring in the reassessments stipulated in the study and also in a questionnaire answered by the patient
% reduction in fat layer assessed by ultrasound, adipometer and photography | Immediately after the procedure and 6 and 20 weeks after
  Adipometer: to measure the thickest point within the treatment area. For the evaluation in the abdominal region, reference points located 5 cm to the side of the umbilical scar, both on the right and left sides, will be recorded. For the evaluation in the flank region, the measurement will be standardized using the axillary midline, being performed exactly in the central fold of each flank; Ultrasound: subcutaneous tissue between the anatomical planes. The probe will be positioned at the points previously marked in the treatment area, following the same measurement performed for adipometry; Photography: at fixed angles and postures with standardized disposable underwear. Three-dimensional images will be taken of the subjects in sagittal (left and right sides) and coronal (front and back sides) views at baseline and at the stipulated follow-up periods. The abdominal region will be exposed and the subject will be instructed to remain still while the camera captures an image.

SECONDARY OUTCOMES:
Patient"s satisfaction assessed by GAIS scale | 6 weeks and 20 weeks after the cryolipolysis procedure
  Patient satisfaction level will be categorized using the 5-point Global Aesthetic Improvement Scale (GAIS). It is divided into 5: "excellent", 4: "greatly improved", 3: "improved", 2: "no change" and 1: "worsened".

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - UNDB, São Luís, Maranhão
  - Clinica Franciele Doneda Estetica Integrada, Paranavaí, Paraná
  - UNIFAE, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Faulhaber J, Sandhofer M, Weiss C, Sattler G, Sadick NS. Effective noninvasive body contouring by using a combination of cryolipolysis, injection lipolysis, and shock waves. J Cosmet Dermatol. 2019 Aug;18(4):1014-1019. doi: 10.1111/jocd.12953. Epub 2019 Apr 13. PMID 30980602
- [Background] Falster M, Schardong J, Santos DPD, Machado BC, Peres A, Rosa PVD, Plentz RDM. Effects of cryolipolysis on lower abdomen fat thickness of healthy women and patient satisfaction: a randomized controlled trial. Braz J Phys Ther. 2020 Sep-Oct;24(5):441-448. doi: 10.1016/j.bjpt.2019.07.005. Epub 2019 Jul 26. PMID 31375459
- [Background] Dierickx CC, Mazer JM, Sand M, Koenig S, Arigon V. Safety, tolerance, and patient satisfaction with noninvasive cryolipolysis. Dermatol Surg. 2013 Aug;39(8):1209-16. doi: 10.1111/dsu.12238. Epub 2013 May 2. PMID 23639062
- [Background] Coleman SR, Sachdeva K, Egbert BM, Preciado J, Allison J. Clinical efficacy of noninvasive cryolipolysis and its effects on peripheral nerves. Aesthetic Plast Surg. 2009 Jul;33(4):482-8. doi: 10.1007/s00266-008-9286-8. Epub 2009 Mar 19. PMID 19296153
- [Background] Boey GE, Wasilenchuk JL. Fat reduction in the inner thigh using a prototype cryolipolysis applicator. Dermatol Surg. 2014 Sep;40(9):1004-9. doi: 10.1097/01.DSS.0000452628.99209.4f. PMID 25111437
- [Background] Bernstein EF, Bloom JD, Basilavecchio LD, Plugis JM. Non-invasive fat reduction of the flanks using a new cryolipolysis applicator and overlapping, two-cycle treatments. Lasers Surg Med. 2014 Dec;46(10):731-5. doi: 10.1002/lsm.22302. Epub 2014 Nov 13. PMID 25395266
- [Background] Bernstein EF, Bloom JD. Safety and Efficacy of Bilateral Submental Cryolipolysis With Quantified 3-Dimensional Imaging of Fat Reduction and Skin Tightening. JAMA Facial Plast Surg. 2017 Sep 1;19(5):350-357. doi: 10.1001/jamafacial.2017.0102. PMID 28426847
- [Background] Abdel-Aal NM, Elerian AE, Elmakaky AM, Alhamaky DMA. Systemic Effects of Cryolipolysis in Central Obese Women: A Randomized Controlled Trial. Lasers Surg Med. 2020 Dec;52(10):971-978. doi: 10.1002/lsm.23250. Epub 2020 Apr 15. PMID 32293044